CLINICAL TRIAL: NCT06131775
Title: Characterisation of TLR4+ Blood Cells in Patients With Solid Cancer
Acronym: ODYSSEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL23_0596; 2023-A01542-43 (Other: ID-RCB)
Record Dates: First submitted 2023-10-13; First posted 2023-11-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: All Types of Solid Cancer
Keywords: Immunotherapy; Innate immune system systemic activation; TLR4 positive immune cells; Lipopolysaccharides; Immunostimulant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunotherapy (Other): Patients with locally advanced/metastatic disease who are due to receive as a first attempt an immune checkpoint inhibitors immunotherapy-based treatment.
  Blood sample collection : One blood draw of 10 mL will be realized before the initiation of immunotherapy. Any adverse event related to the blood draw will be recorded. A follow-up will be performed at 6 months to record the immune-related adverse events, a statement of the disease and any other cancer treatments received. A 24 months long term follow up will be performed to record patient vital status and any date of disease progression.
  Interventions: Biological: Blood sampling
- Curative surgery (Other): Patients newly diagnosed and naive of any anticancer treatment who are due to receive a curative surgery of their primitive tumor.
  Blood samples collection : Three blood draws of 10 mL will be realized : one before the surgery, one after 3 months and one after 6 months. Any adverse event related to the blood draw will be recorded. A follow-up will be performed at 6 months to record the statement of the disease and any other cancer treatments received. A 24 months long term follow up will be performed to record patient vital status and any date of disease relapse.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — One blood sample of 10mL is realized before initiation of immunotherapy
  Arms: Immunotherapy
Biological: Blood sampling — Three blood samples of 10mL are realized at distinct steps of patients disease management : one before the curative surgery, one after three months and one after six months.
  Arms: Curative surgery

SUMMARY:
The potential of immunotherapy in the treatment of cancer is now well documented. While excessive activation of the immune system may be associated with severe reactions and/or auto-immune syndromes, it is now clearly established that controlled activation of the adaptive immune system constitutes a major contribution to the treatment of cancer. Antigen-independent activation of the adaptative immune system with " immune checkpoint inhibitors " (ICI) has allowed prolonged survival in a minority of patients with previously intractable disease. However, a variety of tumor indications are still presently inaccessible to immunotherapeutic approaches or poorly responsive to these therapies.

The immune system is a highly reactive complex comprising antigen-specific cells (adaptive immune system) and antigen-agnostic cells (innate immune system) which interact closely in a complex network. The adaptive immune response is mediated by B and T cells upon antigen-specific recognition. The innate response is mediated by macrophages, dendritic cells, Natural Killer cells and assume the immediate defense of the organism against infectious agents. The innate immune system plays a key role in antigen processing and presentation, production of key cytokines and as anti-tumor effector cells. The role of the innate immune system in the control of cancer progression and in cancer therapy is well documented. Natural Killer cells, involved in antibody-dependent cellular cytotoxicity, and cells performing phagocytosis such as macrophages and neutrophils, participate in tumor destruction after intervention of adaptive immune cells and in combination with certain tumor-targeting therapies, such as antibodies recognizing tumor-specific antigens.

The Odyssey project aims to harness the next generation paradigm of cancer immunotherapy : systemic stimulation of the innate immune system.

To achieve this endeavour the investigator will exploit a well-known yet poorly documented phenomenon, i.e. the rare occurrence of cure in cancer patients who have presented a simultaneous severe septic episode at the time of diagnosis.

Several clinical studies have been realized in order to demonstrate the effect of the innate immune response activation by the bacterial LPS (lipopolysaccharides) in cancer therapy. However, severe toxicities have been described even at very low dose of LPS. The LPS-activated immune response is mediated by TLR4 (Toll Like Receptor 4), a transmembrane receptor expressed by several cell types including monocytes and macrophages. The interaction of TLR4 with LPS mainly induces the release of proinflammatory cytokines (so called " canonical pathway "). TLR4-signalling cascade can also induce the release of type I interferon (so called " alternative pathway "), a class of cytokines known to promote antitumoral activity. LPS tolerance is presumed to be rather associated with the activation of the alternative pathway. Therefore, managing this LPS tolerance is a key mechanism that could limit the systemic toxicity of LPS while stimulating the innate immune system.

Héphaïstos-Pharma biotech and the CRCL Onco-Pharmacology lab (Centre de Recherche en Cancérologie de Lyon) have set up a modified formulation of the LPS that improves its pharmacokinetic properties, reduces its toxicity, and preferentially activates TLR4-alternative signalling pathway. Before investigating the effect of this new immunostimulant in a future phase I/II clinical trial, a translational study is required to further characterize the TLR4 positive cells population as well as the innate immune system in patients with solid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Patient who gave its written informed consent to participate to the study
* Patient with histologically confirmed diagnosis of any type of malignancy (solid tumors)
* Patient with a minimum of 6 months life expectation at inclusion
* Patient covered by a medical insurance

Inclusion criteria specific to cohort 1:

- Patient with metastatic disease or unresectable locally advanced malignancy (solid tumors) who is naive of immune checkpoint inhibitors (ICI)-based immunotherapy and is due to initiate an ICI immunotherapy alone or in combination with any other systemic anticancer treatment.

Inclusion criteria specific to cohort 2:

- Patient with a diagnosed malignancy amenable to surgery with curative intent who is naive of any anticancer treatment

Exclusion Criteria:

* Patient with secondary malignancy unless this malignancy is cured with no evidence of recurrence for at least 5 years.
* Pregnant or breastfeeding woman or expecting to conceive
* Patient who is deprived of liberty due to judicial or administrative decision
* Patient with known psychiatric disorders that would interfere with cooperation with the requirements of the trial
* Patient admitted in a social or sanitary institution for an objective other than the one of this trial
* Adult patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 : 24 months-progression free survival (24M PFS) | 24 months
  Cohort 1 : 24M-PFS defined as the time from the date of the first drug administration to the first documented clinical, biological or radiological progression according to investigator assessment during a period of 24 months. Patients who have not progressed at the time of analysis will be censored at the time of the latest date of assessment.
Cohort 2 : describe the evolution of the percentage of TLR4+ cells in peripheral blood after curative ablation of a cancerous tumour. | Before surgery, after 3 months and after 6 months.
  Number of TLR4 positive cells before curative surgery and after 3 and 6 months.

SECONDARY OUTCOMES:
Overall Survival (OS) Cohorts 1 and 2 | Baseline,date of death, last recorded date or 24 months
  OS defined as the time from the date of the day of the treatment to the date of death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Concentration of innate and adaptive immune cell population Cohorts 1 and 2 | Baseline
  Concentration of innate and adaptive immune memory cells in peripheral blood as defined by the expression level of specific immunophenotypic cell surface receptors
LPS-mediated activation of TLR4 positive cells Cohorts 1 and 2 | baseline
  LPS-mediated activation of TLR4 positive cells defined as the expression of the membrane marker CD169
Number of high grade (≥3) immune-related adverse events (irAE) Cohort 1 | Baseline ans 6 month
  Number of high grade (≥3) irAE(s) 6 months after initiation of immunotherapy
24 months-relapse free survival (24M RFS) Cohort 2 | Before surgery, after 3 months, after 6 months and after 24 month
  24M-RFS defined as the time from the date of the surgery to the first documented clinical, biological or radiological progression according to investigator assessment during a period of 24 months. Patients who have not relapsed at the time of analysis will be censored at the time of the latest date of assessment.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Pneumology Unit, Bron
  - Dermatology Unit, Pierre-Bénite
  - Oncological and Gynecological Surgery Unit,, Pierre-Bénite
  - Oncology Unit, Hospices Civils de Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No